CLINICAL TRIAL: NCT05220722
Title: A Phase 1b/2 Pressure Enabled Regional Immuno-Oncology Study of Hepatic Arterial Infusion of SD-101 With Systemic Checkpoint Blockade for Hepatocellular Carcinoma and Intrahepatic Cholangiocarcinoma
Brief Title: Pressure Enabled Delivery of SD-101 With Checkpoint Blockade for Primary Liver Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The decision was made to terminate the study after the completion of Phase 1b enrollment and not proceed with Phase 2. Trial termination was not due to patient safety or data concerns.
Sponsor: TriSalus Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TS-PERIO-02
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Hepatocellular Carcinoma; Intrahepatic Cholangiocarcinoma
Keywords: Liver Tumors; SD-101; TLR9 Agonist; HCC; ICC
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma | interventions — pembrolizumab; Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: Phase 1b: Escalating doses of SD-101 will be administered alone (Cohort A), together with pembrolizumab (Cohort B), or together with combined ipilimumab and nivolumab. Three weekly doses of SD-101 are delivered over two cycles via HAI using the Pressure Enabled Drug Delivery (PEDD) method of administration.
  Phase 2: Three weekly infusions of SD-101 will be delivered via PEDD/HAI over two cycles at the dose selected from Phase 1b in combination with systemic single- or dual-agent checkpoint blockade.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SD-101 (Experimental): Three weekly doses of SD-101 given over two cycles via HAI using the PEDD method of administration.
  Interventions: Drug: SD-101; Biological: Pembrolizumab; Biological: Nivolumab; Biological: Ipilimumab

INTERVENTIONS:
Drug: SD-101 — SD-101 doses will be delivered via HAI using the PEDD method of administration.
Biological: Pembrolizumab — During Phase 1b, Cohort B, pembrolizumab will be administered together with SD-101.
  Other Names: Keytruda
Biological: Nivolumab — During Phase 1b, Cohort C, nivolumab will be administered together with ipilimumab and SD-101.
  Other Names: Opdivo
Biological: Ipilimumab — During Phase 1b, Cohort C, ipilimumab will be administered together with nivolumab and SD-101.
  Other Names: Yervoy

SUMMARY:
This is an Open-label, Phase 1b/2 Study of the Pressure-Enabled Hepatic Artery Infusion (HAI) of SD-101, a TLR9 agonist, Alone or in Combination with Intravenous Checkpoint Blockade in Adults with Hepatocellular Carcinoma (HCC) and Intrahepatic Cholangiocarcinoma (ICC).

DETAILED DESCRIPTION:
All patients will receive 2 cycles of SD-101. Each cycle consists of 3 consecutive weekly infusions and Cycles 1 and 2 are separated by one month. Escalating doses of SD-101 will be administered alone (Cohort A), together with pembrolizumab (Cohort B), and together with combined ipilimumab and nivolumab (Cohort C). Cohort B will begin dosing at the minimum anticipated biological effect level (MABEL (2mg SD-101)). Cohort C will begin one dose level below the MTD or optimal dose from Cohort B to optimize safety when adding CPI to SD-101.

Following determination of the recommended MTD or optimal dose of SD-101 and which checkpoint inhibitor (CPI) regimen(s) are tolerated, the study will progress to Phase 2. Patients in Phase 2 will receive the SD-101 dose selected from Phase 1b together with systemic single- or double-agent checkpoint blockade. The choice of single- or double-agent CPI therapy together with SD-101 for Phase 2 will consider safety data in addition to response rates from Cohorts B and C in Phase 1b.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older with locally advanced, metastatic or unresectable hepatocellular carcinoma or intrahepatic cholangiocarcinoma, with the diagnosis confirmed by radiologic, histologic or cytologic analysis or clinical features according to the American Association for the Study of Liver Diseases.
2. Previously received 1 line of standard therapy for liver cancer and with persistent or progressive measurable disease, as defined by RECIST version 1.1, that is not amenable to curative therapies
3. Performance status score of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale (scores range from 0 to 5, with higher numbers reflecting greater disability)
4. Designation of class A to B7 on the Child-Pugh liver function scale (a three-category scale [A, B, or C], with C indicating the most severe compromise of liver function)
5. Adequate hematologic and organ function.
6. Has radiographically, histologically or cytologically confirmed HCC or ICC with liver-only or liver-dominant disease. Liver-dominant will be defined as intrahepatic disease representing the largest fraction of disease.
7. Able to understand the study and provide written informed consent prior to any study procedures
8. Has not received prior cytotoxic chemotherapy, targeted therapy, or external radiation therapy within 14 days prior to C1D1
9. Has not ever received prior embolic HAI therapy with permanent embolic material.

   Note: Previous embolic HAI therapy with permanent embolic material will not be exclusionary if following this therapy, the target vessels are not occluded, and tumors are perfused based on the patient's screening imaging.

   Prior surgical resection or radiofrequency ablation of oligometastatic liver disease is allowed. Liver lesions that received ablative therapies should not be considered target lesions unless they have clearly progressed since the therapy or have viable tumor on contrast enhanced MRI or CT.
10. Has no prior history of or other concurrent malignancy unless the malignancy is clinically insignificant, no ongoing treatment is required, and the patient is clinically stable
11. Has measurable disease in the liver according to RECIST v.1.1 criteria
12. Has a life expectancy of >3 months at screening as estimated by the investigator
13. Has a QTc interval ≤480 msec
14. All associated clinically significant (in the judgment of the investigator) drug-related toxicity from previous cancer therapy must be resolved (to Grade ≤1 or the patient's pretreatment level) prior to study treatment administration (Grade 2 alopecia and endocrinopathies controlled on replacement therapy are allowed).
15. Has adequate organ function at screening as evidenced by:

    * Platelet count >80,000/μL
    * Hemoglobin ≥8.0 g/dL
    * White blood cell count (WBC) >2,000/μL
    * Serum creatinine ≤2.0 mg/dL unless the measured creatinine clearance is ≥30 mL/min calculated by Cockcroft-Gault formula.
    * Total and direct bilirubin ≤2.0 × the upper limit of normal (ULN) and alkaline phosphatase ≤5 × ULN. For patients with documented Gilbert's disease, total bilirubin up to 3.0 mg/dL is allowed.
    * ALT and AST ≤5 × ULN
    * Prothrombin time/International Normalized Ratio (INR) or activated partial thromboplastin time (aPTT) test results at screening ≤1.5 × ULN (this applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose for at least 4 weeks prior to the first dose of study intervention) Note: Laboratory tests with exclusionary results judged by the investigator as not compatible with the patient's clinical status may be repeated once for eligibility purposes.
16. Females of childbearing potential must be nonpregnant and nonlactating, or post-menopausal, and have a negative serum human chorionic gonadotropin (hCG) pregnancy test result at screening and a negative urine or serum pregnancy test prior to the first dose of study intervention.

    * Females of childbearing potential must agree to abstain from sexual activity with nonsterilized male partners, or if sexually active with a nonsterilized male partner must agree to use highly effective methods of contraception from screening, throughout the study and agree to continue using such precautions for 100 days after the final dose of study intervention.
    * Nonsterilized males who are sexually active with a female of childbearing potential must agree to use effective methods of contraception and avoid sperm donation from Day 1 throughout the study and for 30 days after the final dose of study intervention.
17. For patients with a documented FGFR2 mutation, prior treatment with a FGFR2-targeted agent or refusal of treatment with at least one of these agents must be documented. For patients with a documented IHD1 mutation, prior treatment with an IHD1 targeted agent or refusal of treatment with ivosidenib must be documented.

Exclusion Criteria:

1. Has received chemotherapy or an investigational agent within 14 days (or 5 half-lives, whichever is shorter) before C1D1.
2. Has active, untreated brain metastasis.
3. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
4. Has main portal vein thrombosis, or severe portal hypertension as defined by a history of variceal hemorrhage or active ascites accumulation refractory to medical management
5. Has more than 2/3 parenchymal replacement by tumor of both liver lobes.
6. Has Child-Pugh Class B 8-9 or C cirrhosis.
7. Has experienced a Grade 3 or higher immune-related AE from prior CPI therapy.

   Note: Patients who have experienced a Grade 3 immune-related AE from prior CPI therapy will not be excluded if that AE has since recovered to a Grade 1 for a minimum of 14 days.
8. Is unable to be temporarily removed from chronic anticoagulation therapy.
9. Has a history of bleeding disorders.
10. Has active coronavirus disease 2019 (COVID-19), other severe infection, including a liver infection, within 2 weeks before the first dose of study drug, or uncontrolled human immunodeficiency virus (HIV) infection at screening.
11. Has active, known, or suspected autoimmune disease or immune-mediated disease. Type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis or alopecia) not requiring systemic treatment or conditions not expected to recur in the absence of an external trigger are not exclusionary.
12. Is receiving systemic steroid therapy >10 mg of prednisone daily or equivalent or any other immunosuppressive medication at any dose level. Local steroid therapies (e.g., otic, ophthalmic, intra-articular or inhaled medications) are acceptable.
13. Has significant concurrent or intercurrent illness, psychiatric disorder, or alcohol or chemical dependence that would, in the opinion of the Investigator and/or Medical Monitor, compromise their safety or compliance or interfere with interpretation of the study.
14. Lactating women are excluded from study participation.
15. Has previously received SD-101.
16. Medical history of significant hypersensitivity, severe and unresolved immune-mediated reactions, severe infusion-related reactions, or allergic reaction to TLR9 agonists or CPI agents in the judgment of the investigator.
17. Patients who were enrolled in the Phase 1b portion of the study will not be eligible for enrollment in Phase 2.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Phase 1b: To Determine the Safety of SD-101 Alone, in Combination with Pembrolizumab, and in Combination with Nivolumab and Ipilimumab | 12 months
  As a measure of safety, adverse events will be graded according to CTCAE v5.0.
Phase 1b: To Determine the Maximum Tolerable Dose (MTD) or Optimal Dose of SD-101 alone, in Combination with Pembrolizumab, and in Combination with Nivolumab and Ipilimumab | 12 months
  A standard 3+3 dose-escalation design will be employed to determine the MTD or optimal dose.
Phase 2: To Assess Overall Response Rate (ORR) | 12 months
  As a measure of activity, ORR will be assessed. ORR will be assessed using Response Evaluation Criteria in Solid Tumours (RECIST) v1.1.

SECONDARY OUTCOMES:
Phase 1b: Assess Preliminary Efficacy in Terms of iRECIST for Immune Based Therapeutics | 12 months
  As a measure of activity, iRECIST will be utilized to determine ORR.
Phase 1b: Assess Preliminary Efficacy in Terms of modified RECIST (mRECIST) for Immune Based Therapeutics | 12 months
  As a measure of activity, mRECIST will be utilized to determine ORR.
Phase 1b: Assess Preliminary Efficacy in Terms of RECIST v1.1 for Immune Based Therapeutics | 12 months
  As a measure of activity, RECIST 1.1 will be utilized to determine hepatic-specific response rate (HRR).
Phase 1b: Assess Preliminary Efficacy in Terms of RECIST v1.1 for Immune Based Therapeutics | 12 months
  As a measure of activity, RECIST 1.1 will be utilized to determine overall progression-free survival (PFS).
Phase 1b: Assess Preliminary Efficacy in Terms of RECIST v1.1 for Immune Based Therapeutics | 12 months
  As a measure of activity, RECIST 1.1 will be utilized to determine clinical benefit (complete response [CR] + partial response [PR] + stable disease [SD]).
Phase 2: To Assess Treatment-Emergent Adverse Events of the Chosen MTD or Optimal Dose of SD-101 in Combination with CPI | 6 months
  As a measure of safety, adverse events will be graded according to CTCAE v5.0.
Phase 2: Assess Efficacy in Terms of RECIST v1.1 for Immune Based Therapeutics | 12 months
  As a measure of activity, RECIST 1.1 will be utilized to determine duration of response (DOR).
Phase 2: To Assess Overall Survival (OS) | 12 months
  As a measure of activity, OS will be assessed. The events for the assessment of 12-month OS are death events.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Colorado, Aurora, Colorado
  - Columbia University, New York, New York
  - Rhode Island Hospital, Providence, Rhode Island
  - MD Anderson Cancer Center, Houston, Texas